CLINICAL TRIAL: NCT04331704
Title: Advancing New Computer-based Health Outreach Regarding Sexual Behavior (ANCHORS) Study: UH3 Project
Brief Title: ANCHORS Alcohol & Sexual Health Study: UH3 Project
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB201902818-N; UH3AA026214 (NIH); OCR31862 (Other: OnCore University of Florida); F31AA028751 (NIH)
Record Dates: First submitted 2020-03-27; First posted 2020-04-02 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Alcohol Use, Unspecified; Substance Use; Sex Behavior
MeSH Terms: conditions — Alcohol Drinking; Substance-Related Disorders; Sexual Behavior | interventions — Pre-Exposure Prophylaxis; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Ethanol; Restraint, Physical

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Personalized Information (Experimental): Participants randomized to this condition will complete a web-based questionnaire and then receive personalized information regarding their alcohol use and sexual health behavior. They will complete daily, phone-based IVR monitoring for assessment purposes and receive further personalized information based on their responses.
  Interventions: Drug: PrEP acronym (pre-exposure prophylaxis); Behavioral: Initial Web Survey; Behavioral: Interactive Voice Response (IVR) assessment with personalized information; Behavioral: Personalized information based on web-based survey responses & standardized information
- Educational Information (Active Comparator): Participants randomized to this condition will complete a web-based questionnaire and then receive educational material regarding their alcohol use and sexual health behavior. They will complete daily phone-based IVR monitoring for assessment purposes.
  Interventions: Drug: PrEP acronym (pre-exposure prophylaxis); Behavioral: Initial Web Survey; Behavioral: Interactive Voice Response (IVR) monitoring; Behavioral: Educational material on alcohol and sexual health behavior

INTERVENTIONS:
Drug: PrEP acronym (pre-exposure prophylaxis) — A daily tablet containing 245 mg of tenofovir disoproxil fumarate and 200 mg emtricitabine (Truvada; Gilead Sciences) for up to 30 days.
  Other Names: emtricitabine/tenofovir disoproxil fumarate
Behavioral: Initial Web Survey — Web-based assessment questions regarding alcohol and other substance use and sexual health behaviors
Behavioral: Interactive Voice Response (IVR) monitoring — Daily telephone-based assessment on alcohol and other substance use, sexual health behavior and PrEP taking
  Arms: Educational Information
Behavioral: Educational material on alcohol and sexual health behavior — Educational material to provide information, resources and techniques to enhance awareness regarding alcohol and other substance use, along with sexual health behavior.
  Arms: Educational Information
Behavioral: Interactive Voice Response (IVR) assessment with personalized information — Daily telephone-based assessment on alcohol and other substance use, sexual health behavior and PrEP taking with personalized and information based on daily IVR responses
  Arms: Personalized Information
Behavioral: Personalized information based on web-based survey responses & standardized information — Personalized and information on alcohol use and sexual health behavior based on responses to the web-based survey along with standardized information.
  Arms: Personalized Information

SUMMARY:
80 young adult men will complete an initial survey and receive 1 of 2 types of alcohol and sexual health education and information to encourage prevention of alcohol-related problems, HIV and other sexually transmitted infections (STIs). Participants will then take pre-exposure prophylaxis (PrEP) for HIV prevention and complete a daily 5-minute, telephone-based interactive voice response (IVR) assessment of alcohol/substance use, sexual behavior and PrEP taking for 30 days. Medication will all be active PrEP. There is no placebo control in this study. Follow-up will occur after 30-days and 6-months later.

ELIGIBILITY:
Inclusion Criteria:

* Ability to read and write English
* Consumption of 5 or more drinks per drinks in a day at least once in the past 30-days
* Sexual intercourse with another man without condom use at least once in the past 30 days
* HIV seronegative at medical screening
* Report currently taking PrEP willingness to take PrEP

Exclusion Criteria:

* History of clinically significant withdrawal from alcohol, defined as any one of the following: a) a lifetime history of seizures, delirium, or hallucinations during alcohol withdrawal; b) a Clinical Institute Withdrawal Assessment scale score > 8; c) a report of drinking to avoid withdrawal symptoms in the past 12 months; or d) a lifetime history of medical treatment for withdrawal.
* Self report injection drug use
* DSM-5 criteria for moderate or severe current substance use disorder besides alcohol and nicotine.
* Serious psychiatric symptoms
* Use of medications that interfere with PrEP including diuretics, nephrotoxic drugs, non-steroidal anti-inflammatory drugs, antiretroviral drugs or other drugs that may interfere with tenofovir excretion
* Active hepatitis B infection
* The following medical exclusions: serious or life-threatening conditions; inadequate biochemical, hepatic, hematologic, or pancreatic function according to laboratory testing
* Participant reports currently taking injectable PrEP

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — male sex assigned at birth
Enrollment: 88 (Estimated)
Dates: Start 2021-01-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in quantity of drinks per week | Baseline up to 1 and 6-month follow-up
  Change in self-reported number of alcoholic drinks per week
Change in peak drinking quantity | Baseline up to 1 and 6-month follow-up
  Change in self-reported number of alcoholic drinks consumed on one's peak drinking day in the past 30 days
PrEP levels in blood at end of intervention period | 1-month follow-up
  Determine whether or not participants have therapeutic levels of PrEP in their blood samples
PrEP levels in blood at the end of the follow-up period | 6-month follow-up
  Determine whether or not participants have therapeutic levels of PrEP in their blood samples
PrEP prescription fill with supporting documentation in the intervention period | during the 1-month intervention period
  Observation of whether or not a participant opts to fill a prescription for PrEP in the intervention period based on pharmacy documentation
PrEP prescription fills with supporting documentation during the follow-up period | the 6-month follow-up period
  Observation of prescription fills for PrEP with documentation during the follow-up period based on pharmacy documentation

SECONDARY OUTCOMES:
Reduced alcohol use as a reason for adherence to PrEP | Baseline up to 1 and 6-month follow-up
  Test reductions in alcohol use following the intervention as a possible mechanism underlying relationships between the intervention and adherence to PrEP
Change in perceived risk of HIV as a reason for adherence to PrEP | Baseline up to 1 and 6-month follow-up
  Test increase in Perceived Risk of HIV Scale score following the intervention as a possible mechanism underlying relationships between the intervention and adherence to PrEP
Change in sexual risk behavior as a reason for adherence to PrEP | Baseline up to 1 and 6-month follow-up
  Test reduction in Risk Assessment Battery score following the intervention as a possible mechanism underlying relationships between the intervention and adherence to PrEP
Increased motivation for behavior change as a reason for adherence to PrEP | Baseline up to 1 and 6-month follow-up
  Test increased score on the Contemplation Ladder for motivation to avoid risky sexual health behavior, to take PrEP and to reduce drinking following the intervention as a possible mechanism underlying relationships between the intervention and adherence to PrEP

CONTACTS AND LOCATIONS:
Overall Officials: Robert L. Cook, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No